CLINICAL TRIAL: NCT00980655
Title: A Phase 3, Open-label Trial To Evaluate The Safety, Tolerability, And Immunogenicity Of 13-valent Pneumococcal Conjugate Vaccine Followed By 23-valent Pneumococcal Polysaccharide Vaccine In Recipients Of Allogeneic Hematopoietic Stem Cell Transplant Aged 2 Years And Older
Brief Title: Study to Evaluate 13 Valent Pneumococcal Conjugate Vaccine (13vPnC) Vaccine Followed by 23-valent Pneumococcal Polysaccharide Vaccine (23vPS) Vaccine in Allogeneic Hematopoietic Stem Cell Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Prevention
Other Study IDs: 6115A1-3003; B1851022 (Other: Alias Study Number); 2009-012087-13 (EudraCT Number)
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-11

CONDITIONS: Vaccines, Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: 13vPnC; Biological: 23vPS

INTERVENTIONS:
Biological: 13vPnC — 0.5mL 13vPnC dose will be administered intramuscularly into the left limb at visits 1,2,3 and 5.
  Starting 3-6 months after HSCT 3 doses given at monthly intervals. 4th dose given 6 months after 3rd dose.
Biological: 23vPS — 0.5mL dose of 23vPS will be administered intramuscularly at visit 6. 23vPS given 1 month after 4th dose of 13vPnC.

SUMMARY:
People who have received an allogeneic hematopoetic stem cell transplant (HSCT) are more likely than other people to get ill from a germ called Streptococcus pneumoniae. Most people who have had a stem cell transplant are offered a vaccine called 23-valent pneumococcal polysaccharide vaccine (23vPS) to help protect against this germ. The purpose of this study is to evaluate the immune response in HSCT recipients who receive a 13 valent pneumococcal vaccine (13vPnC) followed by 23vPS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject >=2 years of age.
* Allogeneic HSCT for hematologic disorder.
* Allogeneic HSCT with full myeloablative conditioning or reduced intensity conditioning.
* Allogeneic HSCT approximately 3 to 6 months (91 days to 203 days) before enrollment.
* Stable engraftment (absolute neutrophil count (ANC) >1000/µL; platelet count >50,000/µL).
* Complete hematologic remission of underlying disease with very good partial remission (VGPR) acceptable in the case of lymphoma and myeloma.
* Subject or parent/legal guardian expected to be available for the entire study and can be contacted by telephone.
* Subject or parent/legal guardian must be able to complete an electronic diary (e-diary) and complete all relevant study procedures during study participation.
* Hematological recovery as defined by ANC >1000/µL; platelet count >50,000/µL.
* All female and male subjects who are biologically capable of having children must agree to abstinence or commit to the use of a reliable method of birth control from signing of the ICF until for 3 months after the last vaccination.
* Negative urine pregnancy test for all female subjects of child bearing potential.

Exclusion Criteria:

* Autologous HSCT.
* Receipt of donor lymphocyte infusions during the 28 days preceding enrollment.
* Uncontrolled GVHD that in the opinion of the investigator would prevent the subject from participating in the study.
* Lansky/Karnofsky Score <=60%.
* Receipt of plasma products or immunoglobulins during the 60 days preceding enrollment.
* Receipt of rituximab since HSCT.
* Receipt of chemotherapy for relapse of underlying malignant disease since HSCT.
* Human immunodeficiency virus (HIV) infection.
* Lymphoproliferative disorder since HSCT.
* Chronic illnesses with cardiac, pulmonary, renal, or liver failure that in the opinion of the investigator would prevent the subject participating in the study.
* Vaccination with any licensed or experimental pneumococcal vaccine since HSCT.
* Previous anaphylactic reaction to any vaccine or vaccine-related component.
* Bleeding diathesis or condition associated with prolonged bleeding time that would in the opinion of the investigator contraindicate intramuscular injection.
* Participation in another study with ongoing use of an unlicensed investigational product from 28 days before study enrollment until the end of the study.
* Participation in another study with ongoing use of a licensed investigational product that in the opinion of the investigator would interfere with the evaluation of the study objectives.
* Permanent residence in a nursing home or other residential care facility.
* Pregnant or breastfeeding female subject.
* Subject who is a direct relative (child, grandchild, parent, or grandparent) of study personnel, or is a member of the study personnel.
* Receipt of advanced therapy medicinal products (ATMP) including gene therapy products, somatic cell therapy products, and tissue engineered products at any time before enrollment.
* If information is available, - previous allergic or anaphylactic reaction to any vaccine or vaccine-related component in a stem cell donor.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2010-01-18 (Actual); Primary Completion 2013-05-16 (Actual); Study Completion 2013-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (47):
- United States (9):
  - University of Kentucky, Lexington, Kentucky
  - Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Columbia University Medical Center Research Pharmacy, New York, New York
  - Columbia University Medical Center-Presbyterian Hospital Building, New York, New York
  - Columbia University/Taub Institute Irving Center for Clinical Research, New York, New York
  - New York-Presbyterian Morgan Stanley Children's Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
- Belgium (5):
  - Universitair Ziekenhuis Gent, Belgium
  - Algemeen Ziekenhuis St.-Jan A.V., Bruges
  - Clinical University St Luc, Brussels
  - Universitaire Ziekenhuizen Leuven (UZ) Gasthuisberg, Leuven
  - CHU Liege, Liège
- Canada (2):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
- Czechia (2):
  - Fakultni nemocnice Brno/Interni hematoonkologicka klinika, Bmo
  - Fakultni nemocnice v Motole, Prague
- France (8):
  - Hôpital Jean Minjoz, Besançon
  - Hopital Henri Mondor, Créteil
  - Hôpital Henri Mondor, Pharmacie, Créteil
  - Hôpital Saint Louis, Paris
  - CHRU Robert Debré, Paris
  - Hopital Robert Debre, Paris
  - Hopital Saint-Louis, Paris
  - Hopital Robert Debre - Service Pharmacie, Paris
- Germany (8):
  - Charite Universitaetsmedizin, Berlin
  - Clinical Trial Center North MediGate GmbH, Hamburg
  - Klinik und Poliklinik fuer Paediatrische Haematologie und Onkologie, Hamburg
  - Universitaetsklinikum Hamburg Eppendorf Clinical Trial Center North MediGate GmbH, Hamburg
  - Universitaetsklinikum Hamburg-Eppendorf, Onkologisches Zentrum, Hamburg
  - Universitatsklinikum Jena, Jena
  - "Universitaetsklinikum Muenster,, Münster
  - Universitaetsklinikum Muenster, Münster
- UMC Utrecht, Wilhelmina Kinder Ziekenhuis, Utrecht, Netherlands
- Poland (3):
  - Klinika Hematologii i Transplantologii, Gdansk
  - NZOZ "HIPOKRATES-II" Sp. z o.o., Krakow
  - Klinika Transplantacji Szpiku, Onkologii i Hematologii Dzieciecej, Wroclaw
- Spain (4):
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Infantil Niño Jesús, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Sweden (5):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Karolinska Universitetssjukhuset Huddinge, Huddinge
  - Universitetssjukhuset i Lund, Barnonkologen Avd 64, Lund
  - Karolinska University Hospital Huddinge, Stockholm
  - Akademiska Sjukhuset, Infektionskliniken, Uppsala

REFERENCES:
- [Derived] Cordonnier C, Ljungman P, Juergens C, Maertens J, Selleslag D, Sundaraiyer V, Giardina PC, Clarke K, Gruber WC, Scott DA, Schmoele-Thoma B; 3003 Study Group. Immunogenicity, safety, and tolerability of 13-valent pneumococcal conjugate vaccine followed by 23-valent pneumococcal polysaccharide vaccine in recipients of allogeneic hematopoietic stem cell transplant aged >/=2 years: an open-label study. Clin Infect Dis. 2015 Aug 1;61(3):313-23. doi: 10.1093/cid/civ287. Epub 2015 Apr 13. PMID 25870329

RESULTS

PARTICIPANT FLOW:
Groups:
- 13vPnC, 23vPS (Pediatric Participants): Pediatric participants aged 2 to 17 years received 4 single 0.5 milliliter (mL) doses of 13-valent pneumococcal conjugate vaccine (13vPnC) intramuscular injections followed by single 0.5 mL dose of 23-valent pneumococcal polysaccharide vaccine (23vPS) intramuscular injection. 13vPnC Doses 1 to 3 were administered at 1-month intervals, 13vPnC Dose 4 was administered at 6 months after 13vPnC Dose 3, and 23vPS was administered 1 month after 13vPnC Dose 4.
- 13vPnC, 23vPS (Adult Participants): Adult participants aged 18 years and above received 4 single 0.5 mL doses of 13vPnC intramuscular injections followed by single 0.5 mL dose of 23vPS intramuscular injection. 13vPnC Doses 1 to 3 were administered at 1-month intervals, 13vPnC Dose 4 was administered at 6 months after 13vPnC Dose 3, and 23vPS was administered 1 month after 13vPnC Dose 4.
Period: Overall Study
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants)
Started | 61 | 190
Vaccinated 13vPnC Dose 1 | 59 | 188
Vaccinated 13vPnC Dose 2 | 55 | 176
Vaccinated 13vPnC Dose 3 | 54 | 167
Vaccinated 13vPnC Dose 4 | 46 | 146
Vaccinated 23vPS Dose | 45 | 140
Completed | 45 | 139
Not Completed | 16 | 51
Not completed — Adverse Event | 13 | 31
Not completed — Death | 0 | 7
Not completed — Protocol Violation | 2 | 7
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Parent/legal guardian request | 1 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of investigational product and had safety data available.
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | Total
Number analyzed (Participants) | 59 | 188 | 247
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.3 (4.41) | 47.3 (12.39) | 38.4 (19.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 74 | 100
  Male | 33 | 114 | 147

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Fold Rise (GMFR) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody From Before 13vPnC Dose 1 to 1 Month After 13vPnC Dose 3 in All Participants
Description: GMFR for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) from before 13vPnC Dose 1 to 1 month after 13vPnC Dose 3 were computed using the logarithmically transformed assay results. Confidence interval (CI) for GMFR were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise. GMFRs were calculated using all participants with available data from both before 13vPnC Dose 1 and after 13vPnC Dose 3 blood draws.
Time Frame: Before 13vPnC Dose 1 (pre-vaccination), 1 month after 13vPnC Dose 3
Population: Evaluable immunogenicity population:eligible participants who received vaccination as assigned;had blood drawn within pre-specified time-frames;had at least 1 valid, determinate assay result; had no major protocol violation. N (number of participants analyzed)=participants evaluable for this measure, n=participants evaluable for specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Groups:
- 13vPnC, 23vPS (All Participants): All participants aged 2 years and above received 4 single 0.5 mL doses of 13vPnC intramuscular injections followed by single 0.5 mL dose of 23vPS intramuscular injection. 13vPnC Doses 1 to 3 were administered at 1-month intervals, 13vPnC Dose 4 was administered at 6 months after 13vPnC Dose 3, and 23vPS was administered 1 month after 13vPnC Dose 4.
Arm/Group | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 197
fold rise
  Serotype 1 (n=191) | 17.96 [13.63 to 23.66]
  Serotype 3 (n=192) | 5.07 [3.98 to 6.46]
  Serotype 4 (n=193) | 23.85 [17.61 to 32.30]
  Serotype 5 (n=194) | 2.99 [2.46 to 3.63]
  Serotype 6A (n=195) | 5.35 [4.18 to 6.85]
  Serotype 6B (n=192) | 5.18 [3.99 to 6.74]
  Serotype 7F (n=195) | 10.28 [8.15 to 12.96]
  Serotype 9V (n=196) | 5.76 [4.63 to 7.17]
  Serotype 14 (n=197) | 4.95 [3.72 to 6.58]
  Serotype 18C (n=196) | 8.22 [6.36 to 10.62]
  Serotype 19A (n=196) | 3.90 [3.10 to 4.89]
  Serotype 19F (n=195) | 6.73 [5.15 to 8.78]
  Serotype 23F (n=197) | 8.01 [6.11 to 10.51]

2. Secondary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After 13vPnC Dose 3 in Pediatric, Adult and All Participants
Description: Antibody GMC for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) for pediatric, adult and all participants are presented. GMC (13vPnC) and corresponding 2-sided 95 percent (%) CIs were evaluated. Geometric means were calculated using all participants with available data for 1 month after 13vPnC Dose 3 blood draw. CI for GMC are back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations.
Time Frame: 1 month after 13vPnC Dose 3
Population: Evaluable immunogenicity population. Here 'N' (number of participants analyzed) signifies all participants who were evaluable for this measure and 'n' signifies all participants who were evaluable for specified serotype for each treatment arm, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter (mcg/mL)
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 49 | 149 | 198
microgram per milliliter (mcg/mL)
  Serotype 1 (n=49, 147, 196) | 3.52 [2.38 to 5.19] | 2.05 [1.53 to 2.76] | 2.35 [1.84 to 2.99]
  Serotype 3 (n=49, 147, 196) | 1.60 [1.13 to 2.26] | 0.62 [0.49 to 0.79] | 0.79 [0.64 to 0.97]
  Serotype 4 (n=49, 147, 196) | 4.13 [2.68 to 6.36] | 1.78 [1.35 to 2.34] | 2.20 [1.73 to 2.78]
  Serotype 5 (n=48, 149, 197) | 4.18 [2.95 to 5.91] | 2.00 [1.60 to 2.51] | 2.39 [1.97 to 2.91]
  Serotype 6A (n=49, 148, 197) | 7.61 [5.16 to 11.23] | 3.31 [2.53 to 4.33] | 4.07 [3.25 to 5.11]
  Serotype 6B (n=48, 147, 195) | 6.29 [3.88 to 10.19] | 3.00 [2.25 to 3.98] | 3.60 [2.81 to 4.61]
  Serotype 7F (n=48, 149, 197) | 7.34 [5.12 to 10.53] | 3.92 [3.08 to 5.00] | 4.57 [3.72 to 5.61]
  Serotype 9V (n=49, 149, 198) | 4.17 [3.01 to 5.78] | 2.44 [1.93 to 3.10] | 2.79 [2.29 to 3.40]
  Serotype 14 (n=49, 149, 198) | 6.22 [4.03 to 9.61] | 5.99 [4.35 to 8.26] | 6.05 [4.65 to 7.86]
  Serotype 18C (n=49, 148, 197) | 4.17 [2.90 to 5.98] | 3.04 [2.37 to 3.91] | 3.29 [2.67 to 4.05]
  Serotype 19A (n=49, 148, 197) | 8.26 [5.86 to 11.65] | 4.77 [3.77 to 6.04] | 5.47 [4.49 to 6.67]
  Serotype 19F (n=49, 148, 197) | 5.80 [3.80 to 8.84] | 3.48 [2.69 to 4.50] | 3.95 [3.17 to 4.93]
  Serotype 23F (n=49, 149, 198) | 6.74 [4.12 to 11.05] | 3.87 [2.85 to 5.26] | 4.44 [3.42 to 5.77]

3. Secondary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After 13vPnC Dose 4 in Pediatric, Adult and All Participants
Description: Antibody GMC for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) for pediatric, adult and all participants are presented. GMC (13vPnC) and corresponding 2-sided 95% CIs were evaluated. Geometric means were calculated using all participants with available data for 1 month after 13vPnC Dose 4 blood draw. CI for GMC are back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations.
Time Frame: 1 month after 13vPnC Dose 4
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 38 | 124 | 162
mcg/mL
  Serotype 1 (n=38, 123, 161) | 8.75 [5.64 to 13.59] | 4.67 [3.37 to 6.47] | 5.41 [4.13 to 7.10]
  Serotype 3 (n=38, 123, 161) | 1.23 [0.89 to 1.70] | 0.91 [0.71 to 1.17] | 0.97 [0.79 to 1.20]
  Serotype 4 (n=36, 124, 160) | 8.41 [5.15 to 13.72] | 4.56 [3.31 to 6.27] | 5.23 [3.99 to 6.86]
  Serotype 5 (n=38, 122, 160) | 8.43 [6.07 to 11.70] | 5.57 [4.28 to 7.26] | 6.15 [4.95 to 7.64]
  Serotype 6A (n=37, 122, 159) | 16.33 [10.59 to 25.16] | 12.23 [8.81 to 16.98] | 13.08 [9.99 to 17.13]
  Serotype 6B (n=38, 124, 162) | 18.13 [11.15 to 29.47] | 12.13 [8.63 to 17.06] | 13.33 [10.04 to 17.70]
  Serotype 7F (n=38, 124, 162) | 10.37 [7.36 to 14.61] | 8.26 [6.33 to 10.78] | 8.71 [7.00 to 10.83]
  Serotype 9V (n=37, 124, 161) | 7.78 [5.21 to 11.61] | 5.09 [3.93 to 6.59] | 5.61 [4.50 to 6.98]
  Serotype 14 (n=37, 124, 161) | 16.04 [10.04 to 25.63] | 12.24 [9.09 to 16.47] | 13.02 [10.13 to 16.74]
  Serotype 18C (n=38, 122, 160) | 6.54 [4.04 to 10.59] | 6.69 [5.01 to 8.93] | 6.65 [5.20 to 8.51]
  Serotype 19A (n=37, 124, 161) | 16.94 [11.05 to 25.98] | 12.99 [9.78 to 17.26] | 13.81 [10.88 to 17.52]
  Serotype 19F (n=38, 123, 161) | 19.96 [12.19 to 32.68] | 13.69 [9.93 to 18.88] | 14.96 [11.42 to 19.61]
  Serotype 23F (n=38, 123, 161) | 16.65 [10.73 to 25.82] | 12.68 [8.82 to 18.22] | 13.52 [10.07 to 18.15]

4. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody From Before 13vPnC Dose 1 to 1 Month After 13vPnC Dose 3 in Pediatric and Adult Participants
Description: GMFR for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) from before 13vPnC Dose 1 to 1 month after 13vPnC Dose 3 were computed using the logarithmically transformed assay results. CI for GMFR were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise. GMFRs were calculated using all participants with available data from both before 13vPnC Dose 1 and after 13vPnC Dose 3 blood draws.
Time Frame: Before 13vPnC Dose 1 (pre-vaccination), 1 month after 13vPnC Dose 3
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants)
Number analyzed (Participants) | 49 | 148
fold rise
  Serotype 1 (n=48, 143) | 27.64 [16.75 to 45.62] | 15.54 [11.20 to 21.56]
  Serotype 3 (n=48, 144) | 7.58 [4.74 to 12.13] | 4.43 [3.35 to 5.88]
  Serotype 4 (n=49, 144) | 40.83 [23.84 to 69.95] | 19.86 [13.83 to 28.52]
  Serotype 5 (n=47, 147) | 4.11 [2.86 to 5.90] | 2.70 [2.15 to 3.39]
  Serotype 6A (n=48, 147) | 7.49 [4.79 to 11.72] | 4.79 [3.57 to 6.44]
  Serotype 6B (n=47, 145) | 6.02 [3.79 to 9.55] | 4.94 [3.60 to 6.77]
  Serotype 7F (n=48, 147) | 14.65 [9.63 to 22.28] | 9.15 [6.95 to 12.05]
  Serotype 9V (n=48, 148) | 7.64 [5.40 to 10.82] | 5.26 [4.02 to 6.87]
  Serotype 14 (n=49, 148) | 5.01 [2.83 to 8.86] | 4.92 [3.53 to 6.87]
  Serotype 18C (n=49, 147) | 12.59 [7.84 to 20.21] | 7.13 [5.27 to 9.65]
  Serotype 19A (n=49, 147) | 5.04 [3.38 to 7.51] | 3.58 [2.72 to 4.70]
  Serotype 19F (n=49, 146) | 7.66 [4.67 to 12.57] | 6.44 [4.69 to 8.85]
  Serotype 23F (n=49, 148) | 9.73 [5.79 to 16.34] | 7.52 [5.46 to 10.35]

5. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody From Before 13vPnC Dose 1 to 1 Month After 13vPnC Dose 4 in Pediatric, Adult and All Participants
Description: GMFR for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) from before 13vPnC Dose 1 to 1 month after 13vPnC Dose 4 were computed using the logarithmically transformed assay results. CI for GMFR were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise. GMFRs were calculated using all participants with available data from both before 13vPnC Dose 1 and after 13vPnC Dose 4 blood draws.
Time Frame: Before 13vPnC Dose 1 (pre-vaccination), 1 month after 13vPnC Dose 4
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 38 | 123 | 161
fold rise
  Serotype 1 (n=37, 120, 157) | 70.66 [39.20 to 127.36] | 35.81 [25.06 to 51.18] | 42.03 [30.94 to 57.11]
  Serotype 3 (n=37, 120, 157) | 5.88 [3.25 to 10.61] | 6.41 [4.74 to 8.66] | 6.28 [4.81 to 8.19]
  Serotype 4 (n=36, 121, 157) | 90.31 [48.05 to 169.77] | 47.47 [32.09 to 70.22] | 55.02 [39.39 to 76.85]
  Serotype 5 (n=37, 119, 156) | 7.76 [4.81 to 12.51] | 7.29 [5.32 to 9.99] | 7.40 [5.69 to 9.63]
  Serotype 6A (n=36, 121, 157) | 15.62 [9.63 to 25.34] | 17.02 [11.95 to 24.23] | 16.90 [12.47 to 22.34]
  Serotype 6B (n=37, 122, 159) | 16.90 [9.76 to 29.25] | 20.09 [13.94 to 28.94] | 19.29 [14.22 to 26.18]
  Serotype 7F (n=38, 123, 161) | 19.18 [11.75 to 31.33] | 18.69 [13.70 to 25.50] | 18.81 [14.48 to 24.43]
  Serotype 9V (n=36, 122, 158) | 14.90 [9.55 to 23.25] | 11.13 [8.27 to 14.99] | 11.90 [9.27 to 15.27]
  Serotype 14 (n=37, 123, 160) | 12.61 [6.47 to 24.56] | 9.69 [6.80 to 13.80] | 10.30 [7.55 to 14.03]
  Serotype 18C (n=38, 121, 159) | 21.22 [12.05 to 37.36] | 14.40 [10.17 to 20.41] | 15.80 [11.76 to 21.24]
  Serotype 19A (n=37, 123, 160) | 11.46 [7.22 to 18.20] | 9.52 [6.90 to 13.12] | 9.94 [7.61 to 12.98]
  Serotype 19F (n=38, 120, 158) | 29.31 [16.63 to 51.64] | 25.63 [17.56 to 37.43] | 26.47 [19.31 to 36.29]
  Serotype 23F (n=38, 122, 160) | 25.37 [14.69 to 43.83] | 23.02 [15.63 to 33.92] | 23.56 [17.11 to 32.45]

6. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody From 1 Month After 13vPnC Dose 3 to 1 Month After 13vPnC Dose 4 in Pediatric, Adult and All Participants
Description: GMFR for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) from 1 month after 13vPnC Dose 3 to 1 month after 13vPnC Dose 4 were computed using the logarithmically transformed assay results. CI for GMFR were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise. GMFRs were calculated using all participants with available data from both after 13vPnC Dose 3 and after 13vPnC Dose 4 blood draws.
Time Frame: 1 month after 13vPnC Dose 3, 1 month after 13vPnC Dose 4
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 37 | 121 | 157
fold rise
  Serotype 1 (n=37, 119, 156) | 2.80 [1.99 to 3.95] | 2.16 [1.65 to 2.82] | 2.30 [1.85 to 2.86]
  Serotype 3 (n=37, 119, 156) | 0.88 [0.64 to 1.22] | 1.32 [1.07 to 1.62] | 1.20 [1.01 to 1.43]
  Serotype 4 (n=35, 121, 156) | 2.19 [1.51 to 3.19] | 2.32 [1.88 to 2.86] | 2.29 [1.91 to 2.74]
  Serotype 5 (n=37, 119, 156) | 2.25 [1.74 to 2.93] | 2.43 [1.94 to 3.06] | 2.39 [1.99 to 2.87]
  Serotype 6A (n=36, 119, 155) | 2.36 [1.87 to 2.99] | 3.06 [2.35 to 3.98] | 2.88 [2.34 to 3.55]
  Serotype 6B (n=37, 120, 157) | 2.96 [2.09 to 4.19] | 3.10 [2.44 to 3.95] | 3.07 [2.51 to 3.75]
  Serotype 7F (n=36, 121, 157) | 1.51 [1.08 to 2.11] | 1.83 [1.47 to 2.29] | 1.75 [1.46 to 2.11]
  Serotype 9V (n=36, 121, 157) | 2.08 [1.43 to 3.03] | 1.82 [1.48 to 2.23] | 1.88 [1.57 to 2.24]
  Serotype 14 (n=36, 121, 157) | 2.50 [1.65 to 3.80] | 1.68 [1.32 to 2.13] | 1.84 [1.50 to 2.26]
  Serotype 18C (n=37, 118, 155) | 1.64 [1.24 to 2.16] | 1.87 [1.54 to 2.28] | 1.81 [1.54 to 2.13]
  Serotype 19A (n=36, 121, 157) | 2.25 [1.60 to 3.17] | 2.33 [1.91 to 2.85] | 2.31 [1.95 to 2.74]
  Serotype 19F (n=37, 120, 157) | 3.50 [2.15 to 5.68] | 3.65 [2.90 to 4.59] | 3.61 [2.94 to 4.44]
  Serotype 23F (n=37, 120, 157) | 2.49 [1.72 to 3.61] | 2.59 [2.04 to 3.30] | 2.57 [2.10 to 3.14]

7. Other Pre Specified Outcome: Percentage of Pediatric, Adult and All Participants Reporting Pre-specified Local Reactions: 13vPnC Dose 1
Description: Specific local reactions were prompted for each day, and reported using an electronic diary. Redness and Swelling were scaled as Any (redness present or swelling present); Mild (0.5 to 2.0 centimeters [cm] for participants aged 2 to <12 years and 2.5 to 5.0 cm for participants aged >= 12 years); Moderate (2.5 to 7.0 cm for participants aged 2 to <12 years and 5.5 to 10.0 cm for participants aged >= 12 years); Severe (greater than [>] 7.0 cm for participants aged 2 to <12 years and >10.0 cm for participants aged >= 12 years). Pain at injection site was scaled as Any (pain present); Mild (did not interfere with activity); Moderate (interfered with activity); Severe (prevented daily activity).
Time Frame: Within 14 days after 13vPnC Dose 1
Population: Safety population. Here 'N' (number of participants analyzed) signifies participants with known values for any local reaction and 'n' signifies participants with known values for specified local reaction. Participants may be represented in more than 1 category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 52 | 171 | 223
percentage of participants
  Redness: any (n = 38, 130, 168) | 21.1 [9.6 to 37.3] | 11.5 [6.6 to 18.3] | 13.7 [8.9 to 19.8]
  Redness: mild (n = 38, 130, 168) | 15.8 [6.0 to 31.3] | 10.8 [6.0 to 17.4] | 11.9 [7.4 to 17.8]
  Redness: moderate (n = 37, 128, 165) | 10.8 [3.0 to 25.4] | 1.6 [0.2 to 5.5] | 3.6 [1.3 to 7.7]
  Redness: severe (n = 37, 128, 165) | 0.0 [0.0 to 9.5] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 2.2]
  Swelling: any (n = 40, 130, 170) | 25.0 [12.7 to 41.2] | 11.5 [6.6 to 18.3] | 14.7 [9.7 to 20.9]
  Swelling: mild (n = 39, 130, 169) | 10.3 [2.9 to 24.2] | 10.8 [6.0 to 17.4] | 10.7 [6.4 to 16.3]
  Swelling: moderate (n = 39, 128, 167) | 20.5 [9.3 to 36.5] | 0.8 [0.0 to 4.3] | 5.4 [2.5 to 10.0]
  Swelling: severe (n = 37, 128, 165) | 0.0 [0.0 to 9.5] | 0.8 [0.0 to 4.3] | 0.6 [0.0 to 3.3]
  Pain: any (n = 51, 171, 222) | 78.4 [64.7 to 88.7] | 73.1 [65.8 to 79.6] | 74.3 [68.1 to 79.9]
  Pain: mild (n = 48, 169, 217) | 68.8 [53.7 to 81.3] | 69.8 [62.3 to 76.6] | 69.6 [63.0 to 75.6]
  Pain: moderate (n = 42, 138, 180) | 45.2 [29.8 to 61.3] | 22.5 [15.8 to 30.3] | 27.8 [21.4 to 34.9]
  Pain: severe (n = 37, 129, 166) | 5.4 [0.7 to 18.2] | 2.3 [0.5 to 6.6] | 3.0 [1.0 to 6.9]

8. Other Pre Specified Outcome: Percentage of Pediatric, Adult and All Participants Reporting Pre-specified Local Reactions: 13vPnC Dose 2
Description: as for outcome 7
Time Frame: Within 14 days after 13vPnC Dose 2
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 41 | 157 | 198
percentage of participants
  Redness: any (n = 28, 109, 137) | 42.9 [24.5 to 62.8] | 16.5 [10.1 to 24.8] | 21.9 [15.3 to 29.8]
  Redness: mild (n = 26, 108, 134) | 34.6 [17.2 to 55.7] | 15.7 [9.4 to 24.0] | 19.4 [13.1 to 27.1]
  Redness: moderate (n = 26, 103, 129) | 26.9 [11.6 to 47.8] | 1.9 [0.2 to 6.8] | 7.0 [3.2 to 12.8]
  Redness: severe (n = 24, 103, 127) | 4.2 [0.1 to 21.1] | 1.0 [0.0 to 5.3] | 1.6 [0.2 to 5.6]
  Swelling: any (n = 28, 105, 133) | 35.7 [18.6 to 55.9] | 14.3 [8.2 to 22.5] | 18.8 [12.5 to 26.5]
  Swelling: mild (n = 26, 105, 131) | 15.4 [4.4 to 34.9] | 14.3 [8.2 to 22.5] | 14.5 [9.0 to 21.7]
  Swelling: moderate (n = 26, 102, 128) | 26.9 [11.6 to 47.8] | 0.0 [0.0 to 3.6] | 5.5 [2.2 to 10.9]
  Swelling: severe (n = 24, 102, 126) | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 3.6] | 0.0 [0.0 to 2.9]
  Pain: any (n = 40, 154, 194) | 77.5 [61.5 to 89.2] | 74.7 [67.0 to 81.3] | 75.3 [68.6 to 81.2]
  Pain: mild (n = 36, 148, 184) | 66.7 [49.0 to 81.4] | 70.9 [62.9 to 78.1] | 70.1 [62.9 to 76.6]
  Pain: moderate (n = 32, 116, 148) | 53.1 [34.7 to 70.9] | 27.6 [19.7 to 36.7] | 33.1 [25.6 to 41.3]
  Pain: severe (n = 27, 104, 131) | 14.8 [4.2 to 33.7] | 1.9 [0.2 to 6.8] | 4.6 [1.7 to 9.7]

9. Other Pre Specified Outcome: Percentage of Pediatric, Adult and All Participants Reporting Pre-specified Local Reactions: 13vPnC Dose 3
Description: as for outcome 7
Time Frame: Within 14 days after 13vPnC Dose 3
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 37 | 138 | 175
percentage of participants
  Redness: any (n = 25, 95, 120) | 32.0 [14.9 to 53.5] | 9.5 [4.4 to 17.2] | 14.2 [8.5 to 21.7]
  Redness: mild (n = 24, 94, 118) | 20.8 [7.1 to 42.2] | 8.5 [3.7 to 16.1] | 11.0 [6.0 to 18.1]
  Redness: moderate (n = 24, 93, 117) | 20.8 [7.1 to 42.2] | 1.1 [0.0 to 5.8] | 5.1 [1.9 to 10.8]
  Redness: severe (n = 23, 93, 116) | 4.3 [0.1 to 21.9] | 1.1 [0.0 to 5.8] | 1.7 [0.2 to 6.1]
  Swelling: any (n = 28, 93, 121) | 35.7 [18.6 to 55.9] | 8.6 [3.8 to 16.2] | 14.9 [9.1 to 22.5]
  Swelling: mild (n = 27, 93, 120) | 25.9 [11.1 to 46.3] | 8.6 [3.8 to 16.2] | 12.5 [7.2 to 19.8]
  Swelling: moderate (n = 25, 92, 117) | 20.0 [6.8 to 40.7] | 0.0 [0.0 to 3.9] | 4.3 [1.4 to 9.7]
  Swelling: severe (n = 23, 92, 115) | 4.3 [0.1 to 21.9] | 0.0 [0.0 to 3.9] | 0.9 [0.0 to 4.7]
  Pain: any (n = 37, 138, 175) | 70.3 [53.0 to 84.1] | 73.2 [65.0 to 80.4] | 72.6 [65.3 to 79.0]
  Pain: mild (n = 31, 132, 163) | 64.5 [45.4 to 80.8] | 67.4 [58.7 to 75.3] | 66.9 [59.1 to 74.0]
  Pain: moderate (n = 34, 107, 141) | 38.2 [22.2 to 56.4] | 27.1 [19.0 to 36.6] | 29.8 [22.4 to 38.1]
  Pain: severe (n = 24, 93, 117) | 8.3 [1.0 to 27.0] | 3.2 [0.7 to 9.1] | 4.3 [1.4 to 9.7]

10. Other Pre Specified Outcome: Percentage of Pediatric, Adult and All Participants Reporting Pre-specified Local Reactions: 13vPnC Dose 4
Description: as for outcome 7
Time Frame: Within 14 days after 13vPnC Dose 4
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 35 | 116 | 151
percentage of participants
  Redness: any (n = 21, 79, 100) | 71.4 [47.8 to 88.7] | 22.8 [14.1 to 33.6] | 33.0 [23.9 to 43.1]
  Redness: mild (n = 20, 77, 97) | 50.0 [27.2 to 72.8] | 15.6 [8.3 to 25.6] | 22.7 [14.8 to 32.3]
  Redness: moderate (n = 18, 72, 90) | 50.0 [26.0 to 74.0] | 9.7 [4.0 to 19.0] | 17.8 [10.5 to 27.3]
  Redness: severe (n = 16, 73, 89) | 12.5 [1.6 to 38.3] | 4.1 [0.9 to 11.5] | 5.6 [1.8 to 12.6]
  Swelling: any (n = 27, 81, 108) | 66.7 [46.0 to 83.5] | 28.4 [18.9 to 39.5] | 38.0 [28.8 to 47.8]
  Swelling: mild (n = 21, 79, 100) | 38.1 [18.1 to 61.6] | 21.5 [13.1 to 32.2] | 25.0 [16.9 to 34.7]
  Swelling: moderate (n = 23, 72, 95) | 52.2 [30.6 to 73.2] | 6.9 [2.3 to 15.5] | 17.9 [10.8 to 27.1]
  Swelling: severe (n = 15, 73, 88) | 6.7 [0.2 to 31.9] | 4.1 [0.9 to 11.5] | 4.5 [1.3 to 11.2]
  Pain: any (n = 30, 113, 143) | 86.7 [69.3 to 96.2] | 77.0 [68.1 to 84.4] | 79.0 [71.4 to 85.4]
  Pain: mild (n = 25, 105, 130) | 76.0 [54.9 to 90.6] | 71.4 [61.8 to 79.8] | 72.3 [63.8 to 79.8]
  Pain: moderate (n = 24, 85, 109) | 62.5 [40.6 to 81.2] | 31.8 [22.1 to 42.8] | 38.5 [29.4 to 48.3]
  Pain: severe (n = 16, 74, 90) | 12.5 [1.6 to 38.3] | 5.4 [1.5 to 13.3] | 6.7 [2.5 to 13.9]

11. Other Pre Specified Outcome: Percentage of Pediatric, Adult and All Participants Reporting Pre-specified Systemic Events: 13vPnC Dose 1
Description: Specific systemic events (fever >=38 degrees Celsius [C], fatigue, headache, vomiting, diarrhea, muscle pain, joint pain and use of medication to treat pain/fever) were prompted for each day, and reported using an electronic diary. Fatigue, headache, muscle pain and joint pain were scaled as: Any (symptom present); Mild (did not interfere with activity); Moderate (some interference with activity); Severe (prevented routine daily activity). Vomiting was scaled as: Any (vomiting present); Mild (1-2 times in 24 hours); Moderate (>2 times in 24 hours); Severe (required intravenous hydration). Diarrhea was scaled as: Any (diarrhea present); Mild (2-3 loose stools in 24 hours); Moderate (4-5 loose stools 24 hours); Severe (>=6 loose stools in 24 hours).
Time Frame: Within 14 days after 13vPnC Dose 1
Population: Safety population. Here 'N' (number of participants analyzed) signifies participants with known values for any systemic event and 'n' signifies participants with known values for specified systemic event. Participants may be represented in more than 1 category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 51 | 172 | 223
percentage of participants
  Fever: >=38 degrees C (n = 39, 130, 169) | 12.8 [4.3 to 27.4] | 6.2 [2.7 to 11.8] | 7.7 [4.2 to 12.8]
  Fever: >=38, <38.5 degrees C (n = 37, 130, 167) | 5.4 [0.7 to 18.2] | 6.2 [2.7 to 11.8] | 6.0 [2.9 to 10.7]
  Fever: >=38.5, <39 degrees C (n = 37, 128, 165) | 5.4 [0.7 to 18.2] | 0.0 [0.0 to 2.8] | 1.2 [0.1 to 4.3]
  Fever: >=39, =<40 degrees C (n = 39, 128, 167) | 7.7 [1.6 to 20.9] | 0.0 [0.0 to 2.8] | 1.8 [0.4 to 5.2]
  Fever: >40 degrees C (n = 37, 128, 165) | 0.0 [0.0 to 9.5] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 2.2]
  Fatigue: Any (n = 45, 159, 204) | 53.3 [37.9 to 68.3] | 59.7 [51.7 to 67.4] | 58.3 [51.2 to 65.2]
  Fatigue: Mild (n = 41, 149, 190) | 36.6 [22.1 to 53.1] | 49.0 [40.7 to 57.3] | 46.3 [39.1 to 53.7]
  Fatigue: Moderate (n = 44, 148, 192) | 36.4 [22.4 to 52.2] | 35.8 [28.1 to 44.1] | 35.9 [29.2 to 43.2]
  Fatigue: Severe (n = 37, 136, 173) | 10.8 [3.0 to 25.4] | 11.8 [6.9 to 18.4] | 11.6 [7.2 to 17.3]
  Headache: Any (n = 42, 147, 189) | 45.2 [29.8 to 61.3] | 44.2 [36.0 to 52.6] | 44.4 [37.2 to 51.8]
  Headache: Mild (n = 41, 145, 186) | 39.0 [24.2 to 55.5] | 37.9 [30.0 to 46.4] | 38.2 [31.2 to 45.6]
  Headache: Moderate (n = 40, 134, 174) | 20.0 [9.1 to 35.6] | 17.2 [11.2 to 24.6] | 17.8 [12.4 to 24.3]
  Headache: Severe (n = 37, 130, 167) | 2.7 [0.1 to 14.2] | 2.3 [0.5 to 6.6] | 2.4 [0.7 to 6.0]
  Vomiting: Any (n = 39, 134, 173) | 20.5 [9.3 to 36.5] | 20.9 [14.4 to 28.8] | 20.8 [15.0 to 27.6]
  Vomiting: Mild (n = 38, 134, 172) | 18.4 [7.7 to 34.3] | 17.9 [11.8 to 25.5] | 18.0 [12.6 to 24.6]
  Vomiting: Moderate (n = 38, 128, 166) | 2.6 [0.1 to 13.8] | 3.9 [1.3 to 8.9] | 3.6 [1.3 to 7.7]
  Vomiting: Severe (n = 37, 128, 165) | 5.4 [0.7 to 18.2] | 0.0 [0.0 to 2.8] | 1.2 [0.1 to 4.3]
  Diarrhea: Any (n = 44, 145, 189) | 31.8 [18.6 to 47.6] | 35.9 [28.1 to 44.2] | 34.9 [28.1 to 42.2]
  Diarrhea: Mild (n = 44, 142, 186) | 31.8 [18.6 to 47.6] | 33.8 [26.1 to 42.2] | 33.3 [26.6 to 40.6]
  Diarrhea: Moderate (n = 38, 133, 171) | 5.3 [0.6 to 17.7] | 9.0 [4.7 to 15.2] | 8.2 [4.5 to 13.4]
  Diarrhea: Severe (n = 37, 131, 168) | 0.0 [0.0 to 9.5] | 3.8 [1.3 to 8.7] | 3.0 [1.0 to 6.8]
  Muscle Pain: Any (n = 47, 154, 201) | 55.3 [40.1 to 69.8] | 50.0 [41.8 to 58.2] | 51.2 [44.1 to 58.3]
  Muscle Pain: Mild (n = 43, 148, 191) | 46.5 [31.2 to 62.3] | 42.6 [34.5 to 51.0] | 43.5 [36.3 to 50.8]
  Muscle Pain: Moderate (n = 44, 139, 183) | 36.4 [22.4 to 52.2] | 21.6 [15.1 to 29.4] | 25.1 [19.0 to 32.1]
  Muscle Pain: Severe (n = 37, 131, 168) | 5.4 [0.7 to 18.2] | 5.3 [2.2 to 10.7] | 5.4 [2.5 to 9.9]
  Joint Pain: Any (n = 38, 143, 181) | 26.3 [13.4 to 43.1] | 26.6 [19.5 to 34.6] | 26.5 [20.2 to 33.6]
  Joint Pain: Mild (n = 37, 139, 176) | 18.9 [8.0 to 35.2] | 19.4 [13.2 to 27.0] | 19.3 [13.8 to 25.9]
  Joint Pain: Moderate (n = 38, 137, 175) | 15.8 [6.0 to 31.3] | 14.6 [9.2 to 21.6] | 14.9 [9.9 to 21.0]
  Joint Pain: Severe (n = 37, 130, 167) | 2.7 [0.1 to 14.2] | 3.1 [0.8 to 7.7] | 3.0 [1.0 to 6.8]
  Use of Medication to Treat Pain (n= 40, 136, 176) | 25.0 [12.7 to 41.2] | 13.2 [8.0 to 20.1] | 15.9 [10.8 to 22.2]
  Use of Medication to Treat Fever (n= 41, 133, 174) | 24.4 [12.4 to 40.3] | 14.3 [8.8 to 21.4] | 16.7 [11.5 to 23.1]

12. Other Pre Specified Outcome: Percentage of Pediatric, Adult and All Participants Reporting Pre-specified Systemic Events: 13vPnC Dose 2
Description: as for outcome 11
Time Frame: Within 14 days after 13vPnC Dose 2
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 45 | 146 | 191
percentage of participants
  Fever: >=38 degrees C (n = 26, 105, 131) | 23.1 [9.0 to 43.6] | 6.7 [2.7 to 13.3] | 9.9 [5.4 to 16.4]
  Fever: >=38, <38.5 degrees C (n = 26, 105, 131) | 19.2 [6.6 to 39.4] | 5.7 [2.1 to 12.0] | 8.4 [4.3 to 14.5]
  Fever: >=38.5, <39 degrees C (n = 24, 102, 126) | 8.3 [1.0 to 27.0] | 1.0 [0.0 to 5.3] | 2.4 [0.5 to 6.8]
  Fever: >=39, =<40 degrees C (n = 24, 102, 126) | 8.3 [1.0 to 27.0] | 1.0 [0.0 to 5.3] | 2.4 [0.5 to 6.8]
  Fever: >40 degrees C (n = 24, 102, 126) | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 3.6] | 0.0 [0.0 to 2.9]
  Fatigue: Any (n = 38, 133, 171) | 60.5 [43.4 to 76.0] | 56.4 [47.5 to 65.0] | 57.3 [49.5 to 64.8]
  Fatigue: Mild (n = 31, 125, 156) | 45.2 [27.3 to 64.0] | 39.2 [30.6 to 48.3] | 40.4 [32.6 to 48.5]
  Fatigue: Moderate (n = 33, 122, 155) | 45.5 [28.1 to 63.6] | 37.7 [29.1 to 46.9] | 39.4 [31.6 to 47.5]
  Fatigue: Severe (n = 24, 107, 131) | 12.5 [2.7 to 32.4] | 9.3 [4.6 to 16.5] | 9.9 [5.4 to 16.4]
  Headache: Any (n = 31, 121,152) | 32.3 [16.7 to 51.4] | 35.5 [27.0 to 44.8] | 34.9 [27.3 to 43.0]
  Headache: Mild (n = 30, 117, 147) | 30.0 [14.7 to 49.4] | 29.9 [21.8 to 39.1] | 29.9 [22.7 to 38.0]
  Headache: Moderate (n = 26, 110, 136) | 7.7 [0.9 to 25.1] | 16.4 [10.0 to 24.6] | 14.7 [9.2 to 21.8]
  Headache: Severe (n = 24, 104, 128) | 0.0 [0.0 to 14.2] | 1.9 [0.2 to 6.8] | 1.6 [0.2 to 5.5]
  Vomiting: Any (n = 28, 107, 135) | 21.4 [8.3 to 41.0] | 13.1 [7.3 to 21.0] | 14.8 [9.3 to 21.9]
  Vomiting: Mild (n = 27, 107, 134) | 18.5 [6.3 to 38.1] | 10.3 [5.2 to 17.7] | 11.9 [7.0 to 18.7]
  Vomiting: Moderate (n = 28, 103, 131) | 14.3 [4.0 to 32.7] | 4.9 [1.6 to 11.0] | 6.9 [3.2 to 12.6]
  Vomiting: Severe (n = 24, 102, 126) | 0.0 [0.0 to 14.2] | 1.0 [0.0 to 5.3] | 0.8 [0.0 to 4.3]
  Diarrhea: Any (n = 29, 121, 150) | 31.0 [15.3 to 50.8] | 28.9 [21.0 to 37.9] | 29.3 [22.2 to 37.3]
  Diarrhea: Mild (n = 29, 120, 149) | 31.0 [15.3 to 50.8] | 26.7 [19.0 to 35.5] | 27.5 [20.5 to 35.4]
  Diarrhea: Moderate (n = 25, 109, 134) | 8.0 [1.0 to 26.0] | 10.1 [5.1 to 17.3] | 9.7 [5.3 to 16.0]
  Diarrhea: Severe (n = 24, 103, 127) | 0.0 [0.0 to 14.2] | 1.9 [0.2 to 6.8] | 1.6 [0.2 to 5.6]
  Muscle Pain: Any (n = 36, 124, 160) | 44.4 [27.9 to 61.9] | 45.2 [36.2 to 54.3] | 45.0 [37.1 to 53.1]
  Muscle Pain: Mild (n = 32, 118, 150) | 31.3 [16.1 to 50.0] | 37.3 [28.6 to 46.7] | 36.0 [28.3 to 44.2]
  Muscle Pain: Moderate (n = 32, 111, 143) | 37.5 [21.1 to 56.3] | 25.2 [17.5 to 34.4] | 28.0 [20.8 to 36.1]
  Muscle Pain: Severe (n = 25, 106, 131) | 8.0 [1.0 to 26.0] | 5.7 [2.1 to 11.9] | 6.1 [2.7 to 11.7]
  Joint Pain: Any (n = 31, 116, 147) | 32.3 [16.7 to 51.4] | 23.3 [15.9 to 32.0] | 25.2 [18.4 to 33.0]
  Joint Pain: Mild (n = 27, 115, 142) | 18.5 [6.3 to 38.1] | 21.7 [14.6 to 30.4] | 21.1 [14.7 to 28.8]
  Joint Pain: Moderate (n = 30, 106, 136) | 30.0 [14.7 to 49.4] | 10.4 [5.3 to 17.8] | 14.7 [9.2 to 21.8]
  Joint Pain: Severe (n = 25, 104, 129) | 4.0 [0.1 to 20.4] | 1.9 [0.2 to 6.8] | 2.3 [0.5 to 6.6]
  Use of Medication to Treat Pain (n= 28, 105, 133) | 25.0 [10.7 to 44.9] | 7.6 [3.3 to 14.5] | 11.3 [6.5 to 17.9]
  Use of Medication to Treat Fever (n= 27, 107, 134) | 33.3 [16.5 to 54.0] | 10.3 [5.2 to 17.7] | 14.9 [9.4 to 22.1]

13. Other Pre Specified Outcome: Percentage of Pediatric, Adult and All Participants Reporting Pre-specified Systemic Events: 13vPnC Dose 3
Description: as for outcome 11
Time Frame: Within 14 days after 13vPnC Dose 3
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 42 | 136 | 178
percentage of participants
  Fever: >=38 degrees C (n = 27, 93, 120) | 14.8 [4.2 to 33.7] | 4.3 [1.2 to 10.6] | 6.7 [2.9 to 12.7]
  Fever: >=38, <38.5 degrees C (n = 26, 93, 119) | 11.5 [2.4 to 30.2] | 3.2 [0.7 to 9.1] | 5.0 [1.9 to 10.7]
  Fever: >=38.5, <39 degrees C (n = 24, 93, 117) | 4.2 [0.1 to 21.1] | 3.2 [0.7 to 9.1] | 3.4 [0.9 to 8.5]
  Fever: >=39, =<40 degrees C (n = 24, 92, 116) | 4.2 [0.1 to 21.1] | 1.1 [0.0 to 5.9] | 1.7 [0.2 to 6.1]
  Fever: >40 degrees C (n = 23, 92, 115) | 0.0 [0.0 to 14.8] | 0.0 [0.0 to 3.9] | 0.0 [0.0 to 3.2]
  Fatigue: Any (n = 35, 122, 157) | 48.6 [31.4 to 66.0] | 49.2 [40.0 to 58.4] | 49.0 [41.0 to 57.1]
  Fatigue: Mild (n = 32, 116, 148) | 40.6 [23.7 to 59.4] | 38.8 [29.9 to 48.3] | 39.2 [31.3 to 47.5]
  Fatigue: Moderate (n = 30, 107, 137) | 33.3 [17.3 to 52.8] | 29.9 [21.4 to 39.5] | 30.7 [23.1 to 39.1]
  Fatigue: Severe (n = 24, 96, 120) | 4.2 [0.1 to 21.1] | 7.3 [3.0 to 14.4] | 6.7 [2.9 to 12.7]
  Headache: Any (n = 32, 110,142) | 37.5 [21.1 to 56.3] | 37.3 [28.2 to 47.0] | 37.3 [29.4 to 45.8]
  Headache: Mild (n = 30, 108, 138) | 30.0 [14.7 to 49.4] | 32.4 [23.7 to 42.1] | 31.9 [24.2 to 40.4]
  Headache: Moderate (n = 27, 95, 122) | 22.2 [8.6 to 42.3] | 15.8 [9.1 to 24.7] | 17.2 [11.0 to 25.1]
  Headache: Severe (n = 25, 94, 119) | 8.0 [1.0 to 26.0] | 2.1 [0.3 to 7.5] | 3.4 [0.9 to 8.4]
  Vomiting: Any (n = 25, 95, 120) | 8.0 [1.0 to 26.0] | 11.6 [5.9 to 19.8] | 10.8 [5.9 to 17.8]
  Vomiting: Mild (n = 24, 95, 119) | 4.2 [0.1 to 21.1] | 5.3 [1.7 to 11.9] | 5.0 [1.9 to 10.7]
  Vomiting: Moderate (n = 24, 93, 117) | 4.2 [0.1 to 21.1] | 7.5 [3.1 to 14.9] | 6.8 [3.0 to 13.0]
  Vomiting: Severe (n = 23, 92, 115) | 0.0 [0.0 to 14.8] | 0.0 [0.0 to 3.9] | 0.0 [0.0 to 3.2]
  Diarrhea: Any (n = 26, 104, 130) | 15.4 [4.4 to 34.9] | 25.0 [17.0 to 34.4] | 23.1 [16.1 to 31.3]
  Diarrhea: Mild (n = 26, 102, 128) | 15.4 [4.4 to 34.9] | 21.6 [14.0 to 30.8] | 20.3 [13.7 to 28.3]
  Diarrhea: Moderate (n = 24, 95, 119) | 4.2 [0.1 to 21.1] | 5.3 [1.7 to 11.9] | 5.0 [1.9 to 10.7]
  Diarrhea: Severe (n = 23, 94, 117) | 0.0 [0.0 to 14.8] | 2.1 [0.3 to 7.5] | 1.7 [0.2 to 6.0]
  Muscle Pain: Any (n = 35, 117, 152) | 45.7 [28.8 to 63.4] | 38.5 [29.6 to 47.9] | 40.1 [32.3 to 48.4]
  Muscle Pain: Mild (n = 30, 112, 142) | 33.3 [17.3 to 52.8] | 33.0 [24.4 to 42.6] | 33.1 [25.4 to 41.5]
  Muscle Pain: Moderate (n = 31, 101, 132) | 32.3 [16.7 to 51.4] | 16.8 [10.1 to 25.6] | 20.5 [13.9 to 28.3]
  Muscle Pain: Severe (n = 24, 94, 118) | 4.2 [0.1 to 21.1] | 3.2 [0.7 to 9.0] | 3.4 [0.9 to 8.5]
  Joint Pain: Any (n = 28, 104, 132) | 25.0 [10.7 to 44.9] | 20.2 [13.0 to 29.2] | 21.2 [14.6 to 29.2]
  Joint Pain: Mild (n = 26, 102, 128) | 19.2 [6.6 to 39.4] | 17.6 [10.8 to 26.4] | 18.0 [11.7 to 25.7]
  Joint Pain: Moderate (n = 27, 95, 122) | 18.5 [6.3 to 38.1] | 8.4 [3.7 to 15.9] | 10.7 [5.8 to 17.5]
  Joint Pain: Severe (n = 25, 94, 119) | 8.0 [1.0 to 26.0] | 2.1 [0.3 to 7.5] | 3.4 [0.9 to 8.4]
  Use of Medication to Treat Pain (n= 28, 97, 125) | 21.4 [8.3 to 41.0] | 12.4 [6.6 to 20.6] | 14.4 [8.8 to 21.8]
  Use of Medication to Treat Fever (n= 30, 101, 131) | 26.7 [12.3 to 45.9] | 15.8 [9.3 to 24.4] | 18.3 [12.1 to 26.0]

14. Other Pre Specified Outcome: Percentage of Pediatric, Adult and All Participants Reporting Pre-specified Systemic Events: 13vPnC Dose 4
Description: as for outcome 11
Time Frame: Within 14 days after 13vPnC Dose 4
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC, 23vPS (Pediatric Participants) | 13vPnC, 23vPS (Adult Participants) | 13vPnC, 23vPS (All Participants)
Number analyzed (Participants) | 32 | 116 | 148
percentage of participants
  Fever: >=38 degrees C (n= 18, 78, 96) | 27.8 [9.7 to 53.5] | 15.4 [8.2 to 25.3] | 17.7 [10.7 to 26.8]
  Fever: >=38, <38.5 degrees C (n = 16, 76, 92) | 12.5 [1.6 to 38.3] | 13.2 [6.5 to 22.9] | 13.0 [6.9 to 21.7]
  Fever: >=38.5, <39 degrees C (n = 17, 73, 90) | 17.6 [3.8 to 43.4] | 2.7 [0.3 to 9.5] | 5.6 [1.8 to 12.5]
  Fever: >=39, =<40 degrees C (n = 15, 72, 87) | 0.0 [0.0 to 21.8] | 2.8 [0.3 to 9.7] | 2.3 [0.3 to 8.1]
  Fever: >40 degrees C (n = 15, 71, 86) | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 5.1] | 0.0 [0.0 to 4.2]
  Fatigue: Any (n = 28, 100, 128) | 67.9 [47.6 to 84.1] | 67.0 [56.9 to 76.1] | 67.2 [58.3 to 75.2]
  Fatigue: Mild (n = 26, 95, 121) | 61.5 [40.6 to 79.8] | 54.7 [44.2 to 65.0] | 56.2 [46.9 to 65.2]
  Fatigue: Moderate (n = 20, 86, 106) | 45.0 [23.1 to 68.5] | 45.3 [34.6 to 56.5] | 45.3 [35.6 to 55.2]
  Fatigue: Severe (n = 16, 77, 93) | 12.5 [1.6 to 38.3] | 13.0 [6.4 to 22.6] | 12.9 [6.8 to 21.5]
  Headache: Any (n = 21, 93, 114) | 52.4 [29.8 to 74.3] | 45.2 [34.8 to 55.8] | 46.5 [37.1 to 56.1]
  Headache: Mild (n = 21, 88, 109) | 47.6 [25.7 to 70.2] | 38.6 [28.4 to 49.6] | 40.4 [31.1 to 50.2]
  Headache: Moderate (n = 16, 82, 98) | 18.8 [4.0 to 45.6] | 28.0 [18.7 to 39.1] | 26.5 [18.1 to 36.4]
  Headache: Severe (n = 16, 74, 90) | 12.5 [1.6 to 38.3] | 5.4 [1.5 to 13.3] | 6.7 [2.5 to 13.9]
  Vomiting: Any (n = 16, 73, 89) | 6.3 [0.2 to 30.2] | 5.5 [1.5 to 13.4] | 5.6 [1.8 to 12.6]
  Vomiting: Mild (n = 16, 73, 89) | 6.3 [0.2 to 30.2] | 5.5 [1.5 to 13.4] | 5.6 [1.8 to 12.6]
  Vomiting: Moderate (n = 15, 71, 86) | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 5.1] | 0.0 [0.0 to 4.2]
  Vomiting: Severe (n = 15, 71, 86) | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 5.1] | 0.0 [0.0 to 4.2]
  Diarrhea: Any (n = 18, 83, 101) | 22.2 [6.4 to 47.6] | 30.1 [20.5 to 41.2] | 28.7 [20.1 to 38.6]
  Diarrhea: Mild (n = 18, 82, 100) | 22.2 [6.4 to 47.6] | 29.3 [19.7 to 40.4] | 28.0 [19.5 to 37.9]
  Diarrhea: Moderate (n = 15, 72, 87) | 0.0 [0.0 to 21.8] | 4.2 [0.9 to 11.7] | 3.4 [0.7 to 9.7]
  Diarrhea: Severe (n = 15, 72, 87) | 0.0 [0.0 to 21.8] | 1.4 [0.0 to 7.5] | 1.1 [0.0 to 6.2]
  Muscle Pain: Any (n = 24, 99, 123) | 58.3 [36.6 to 77.9] | 60.6 [50.3 to 70.3] | 60.2 [50.9 to 68.9]
  Muscle Pain: Mild (n = 22, 92, 114) | 50.0 [28.2 to 71.8] | 50.0 [39.4 to 60.6] | 50.0 [40.5 to 59.5]
  Muscle Pain: Moderate (n = 19, 80, 99) | 36.8 [16.3 to 61.6] | 30.0 [20.3 to 41.3] | 31.3 [22.4 to 41.4]
  Muscle Pain: Severe (n = 16, 75, 91) | 12.5 [1.6 to 38.3] | 6.7 [2.2 to 14.9] | 7.7 [3.1 to 15.2]
  Joint Pain: Any (n = 16, 83, 99) | 25.0 [7.3 to 52.4] | 32.5 [22.6 to 43.7] | 31.3 [22.4 to 41.4]
  Joint Pain: Mild (n = 15, 78, 93) | 13.3 [1.7 to 40.5] | 24.4 [15.3 to 35.4] | 22.6 [14.6 to 32.4]
  Joint Pain: Moderate (n = 16, 75, 91) | 12.5 [1.6 to 38.3] | 17.3 [9.6 to 27.8] | 16.5 [9.5 to 25.7]
  Joint Pain: Severe (n = 16, 74, 90) | 6.3 [0.2 to 30.2] | 4.1 [0.8 to 11.4] | 4.4 [1.2 to 11.0]
  Use of Medication to Treat Pain (n= 16, 77, 93) | 18.8 [4.0 to 45.6] | 16.9 [9.3 to 27.1] | 17.2 [10.2 to 26.4]
  Use of Medication to Treat Fever (n= 17, 77, 94) | 23.5 [6.8 to 49.9] | 15.6 [8.3 to 25.6] | 17.0 [10.1 to 26.2]

ADVERSE EVENTS:
Time Frame: AEs/SAEs: recorded from 13vPnC Dose 1 to completion of study. Participants recorded pre-specified AEs in electronic diary:local reactions; systemic events (up to 14 days after 13vPnC vaccination)
Description: SAEs and AEs were grouped by system organ class and summarized. AEs included AEs collected in electronic diary (local,systemic reactions for 13vPnC; systematic assessment) and AEs collected on case report form at each visit (nonsystematic assessment). Participants who received specified dose and had safety data available were evaluable for safety.
Groups:
- 13vPnC Dose 1 to 13vPnC Dose 3 Blood Draw: All participants aged 2 years and above who received 3 single 0.5 mL doses of 13vPnC intramuscular injections at 1-month intervals, were assessed from 13vPnC Dose 1 to the blood draw 1 month after 13vPnC Dose 3.
- 13vPnC Dose 3 Blood Draw to 13vPnC Dose 4: All participants aged 2 years and above who received 4 single 0.5 mL doses of 13vPnC intramuscular injections, 13vPnC Doses 1 to 3 at 1-month intervals and 13vPnC Dose 4 at 6 months after 13vPnC Dose 3, were assessed from blood draw 1 month after 13vPnC Dose 3 to prior to administration of 13vPnC Dose 4.
- 13vPnC Dose 4: All participants aged 2 years and above who received 4 single 0.5 mL doses of 13vPnC intramuscular injections, 13vPnC Doses 1 to 3 at 1-month intervals and 13vPnC Dose 4 at 6 months after 13vPnC Dose 3, were assessed from 13vPnC Dose 4 to the blood draw 1 month after 13vPnC Dose 4.
- 23vPS Dose: All participants aged 2 years and above who received 4 single 0.5 mL doses of 13vPnC intramuscular injections, 13vPnC Doses 1 to 3 at 1-month intervals and 13vPnC Dose 4 at 6 months after 13vPnC Dose 3, followed by single 0.5 mL dose of 23vPS intramuscular injection at 1 month after 13vPnC Dose 4, were assessed from 23vPS Dose to the blood draw 1 month after 23vPS Dose.
- Follow-up: All participants aged 2 years and above who received 4 single 0.5 mL doses of 13vPnC intramuscular injections, 13vPnC Doses 1 to 3 at 1-month intervals and 13vPnC Dose 4 at 6 months after 13vPnC Dose 3, followed by single 0.5 mL dose of 23vPS intramuscular injection at 1 month after 13vPnC Dose 4, were assessed from blood draw 1 month after 23vPS Dose to 6-month follow-up.
Arm/Group | 13vPnC Dose 1 to 13vPnC Dose 3 Blood Draw | 13vPnC Dose 3 Blood Draw to 13vPnC Dose 4 | 13vPnC Dose 4 | 23vPS Dose | Follow-up
Serious Adverse Events (participants affected / at risk) | 58/247 | 42/221 | 11/192 | 11/184 | 28/247
Other Adverse Events (participants affected / at risk) | 203/247 | 89/221 | 127/192 | 93/184 | 19/247
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC Dose 1 to 13vPnC Dose 3 Blood Draw (N=247) | 13vPnC Dose 3 Blood Draw to 13vPnC Dose 4 (N=221) | 13vPnC Dose 4 (N=192) | 23vPS Dose (N=184) | Follow-up (N=247)
Haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 0
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Warm type haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Hernial eventration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 6 | 4 | 0 | 0 | 4
Injection site erythema (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 1 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Graft versus host disease (Immune system disorders) | 5 | 1 | 0 | 0 | 2
Graft versus host disease in intestine (Immune system disorders) | 2 | 0 | 0 | 0 | 0
Chronic graft versus host disease (Immune system disorders) | 1 | 0 | 0 | 0 | 1
Graft versus host disease in liver (Immune system disorders) | 1 | 1 | 0 | 2 | 0
Graft versus host disease in skin (Immune system disorders) | 1 | 2 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 2 | 2 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 2 | 4 | 1 | 1 | 2
Pneumonia (Infections and infestations) | 2 | 2 | 1 | 0 | 4
Respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Cerebral toxoplasmosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Enterocolitis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Molluscum contagiosum (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia haemophilus (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Haemophilus sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Hepatic candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Hepatitis B (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes zoster disseminated (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia pseudomonas aeruginosa (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
H1N1 influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Thrombophlebitis septic (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Varicella (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Cytomegalovirus test positive (Investigations) | 0 | 1 | 0 | 0 | 0
False positive investigation result (Investigations) | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2 | 0 | 0 | 0
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 4 | 1 | 0 | 3
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Plasma cell myeloma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Refractory anaemia with an excess of blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Juvenile chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Uncoded (General disorders) | 0 | 1 | 0 | 0 | 1 — Term was not coded because it violated sponsor's coding conventions.
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC Dose 1 to 13vPnC Dose 3 Blood Draw (N=247) | 13vPnC Dose 3 Blood Draw to 13vPnC Dose 4 (N=221) | 13vPnC Dose 4 (N=192) | 23vPS Dose (N=184) | Follow-up (N=247)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 2 | 0 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
Aplasia pure red cell (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Hypergammaglobulinaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Dilatation ventricular (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myotonic dystrophy (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Ichthyosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 3 | 2 | 0 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Ear pruritus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Cushingoid (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 1 | 0 | 0 | 0
Cushing's syndrome (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1 | 0 | 0
Oestrogen deficiency (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 6 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 5 | 3 | 1 | 2 | 0
Allergic keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0 | 0
Foreign body sensation in eyes (Eye disorders) | 1 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 1
Orbital oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 1 | 0
Vitreous detachment (Eye disorders) | 0 | 2 | 0 | 0 | 0
Blindness (Eye disorders) | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0
Eye inflammation (Eye disorders) | 0 | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0 | 0
Xerophthalmia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 24 | 2 | 3 | 3 | 1
Vomiting (Gastrointestinal disorders) | 15 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 0 | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 8 | 1 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 5 | 2 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 2 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0 | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Aptyalism (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oral mucosal discolouration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Tongue coated (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Oral lichen planus (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 15 | 3 | 3 | 5 | 0
Pyrexia (General disorders) | 16 | 5 | 3 | 8 | 1
Oedema peripheral (General disorders) | 12 | 6 | 0 | 2 | 0
Asthenia (General disorders) | 10 | 2 | 1 | 3 | 1
Injection site swelling (General disorders) | 4 | 0 | 3 | 8 | 0
Injection site erythema (General disorders) | 3 | 0 | 4 | 5 | 0
Oedema (General disorders) | 3 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 1 | 0 | 1
Catheter site rash (General disorders) | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 1 | 0
Complication of device removal (General disorders) | 1 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 1 | 0 | 1 | 0 | 0
Feeling hot (General disorders) | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 1 | 1 | 0 | 0
Injection site movement impairment (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 5 | 8 | 0
Medical device complication (General disorders) | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 1 | 0 | 0 | 0
Vaccination site haematoma (General disorders) | 1 | 0 | 1 | 0 | 0
Vaccination site pain (General disorders) | 1 | 0 | 0 | 6 | 0
Vaccination site reaction (General disorders) | 1 | 0 | 0 | 4 | 0
Inflammation (General disorders) | 0 | 1 | 0 | 0 | 0
Spinal pain (General disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 1 | 0
Injection site pruritus (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 1 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0
Vaccination site erythema (General disorders) | 0 | 0 | 0 | 5 | 0
Vaccination site swelling (General disorders) | 0 | 0 | 0 | 4 | 0
Injection site induration (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site inflammation (General disorders) | 0 | 0 | 0 | 1 | 0
Vaccination site oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Vaccination site rash (General disorders) | 0 | 0 | 0 | 1 | 0
Hernia (General disorders) | 0 | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 1 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Graft versus host disease (Immune system disorders) | 21 | 8 | 2 | 4 | 0
Chronic graft versus host disease (Immune system disorders) | 12 | 3 | 0 | 3 | 0
Graft versus host disease in liver (Immune system disorders) | 5 | 1 | 0 | 1 | 0
Graft versus host disease in skin (Immune system disorders) | 4 | 6 | 0 | 0 | 0
Food allergy (Immune system disorders) | 2 | 0 | 1 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 2 | 0 | 0 | 0 | 0
Acute graft versus host disease (Immune system disorders) | 1 | 1 | 0 | 0 | 0
Chronic graft versus host disease in liver (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Graft versus host disease in intestine (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 2 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 28 | 6 | 11 | 9 | 0
Cytomegalovirus infection (Infections and infestations) | 10 | 3 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 10 | 6 | 3 | 3 | 1
Herpes zoster (Infections and infestations) | 8 | 5 | 0 | 1 | 2
Bronchitis (Infections and infestations) | 6 | 3 | 1 | 2 | 1
Sinusitis (Infections and infestations) | 5 | 1 | 0 | 2 | 0
Tonsillitis (Infections and infestations) | 5 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 4 | 2 | 0 | 0 | 1
Oral fungal infection (Infections and infestations) | 4 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 4 | 3 | 0 | 2 | 0
Escherichia infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 2 | 1 | 0 | 3 | 0
Oral herpes (Infections and infestations) | 3 | 4 | 1 | 1 | 0
Candidiasis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Enterobacter sepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 2 | 1 | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 2 | 0 | 1 | 2 | 0
Respiratory syncytial virus infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Adenovirus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Aspergillosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Conjunctivitis viral (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Enterobacter infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Genital infection fungal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 3 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Mycoplasma infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Respiratory moniliasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Systemic candida (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Hepatitis B (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes zoster oticus (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Streptococcal urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Herpes virus infection (Infections and infestations) | 10 | 0 | 1 | 0 | 0
Infected dermal cyst (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Toxoplasmosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Viral rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Injection site cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Trichosporon infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Conjunctival scar (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Drug administration error (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Blood testosterone decreased (Investigations) | 2 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 2 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 1 | 1 | 3 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Human herpes virus 6 serology positive (Investigations) | 1 | 0 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0
Thyroxine decreased (Investigations) | 1 | 0 | 0 | 0 | 1
Serum ferritin increased (Investigations) | 0 | 2 | 1 | 0 | 0
Cystogram (Investigations) | 0 | 1 | 0 | 0 | 0
Ejection fraction abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 1 | 0 | 1 | 1
Fluid retention (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 3 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Folate deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Vitamin K deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Haemochromatosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 6 | 4 | 3 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 2 | 2 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 1 | 0 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1 | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Precursor B-lymphoblastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 13 | 3 | 4 | 3 | 0
Dysgeusia (Nervous system disorders) | 3 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 2 | 0 | 0 | 0
Coordination abnormal (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Migraine with aura (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cranial nerve palsies multiple (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 5 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 1 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 2 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 2 | 0
Polyuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 3 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urethral pain (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Genital discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 2 | 4 | 7 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2 | 3 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 14 | 0 | 2 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 2 | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Generalised erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Lichenification (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0
Perivascular dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Pityriasis rubra pilaris (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 7 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 1 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Vasodilatation (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Venous insufficiency (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Redness (Any) (Skin and subcutaneous tissue disorders) | 23/168 | 0/0 | 33/100 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Redness (Mild) (Skin and subcutaneous tissue disorders) | 20/168 | 0/0 | 22/97 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 6/165 | 0/0 | 16/90 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Redness (Severe) (Skin and subcutaneous tissue disorders) | 0/165 | 0/0 | 5/89 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Swelling (Any) (Skin and subcutaneous tissue disorders) | 25/170 | 0/0 | 41/108 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 18/169 | 0/0 | 25/100 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 9/167 | 0/0 | 17/95 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 1/165 | 0/0 | 4/88 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Pain (Any) (Skin and subcutaneous tissue disorders) | 165/222 | 0/0 | 113/143 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Pain (Mild) (Skin and subcutaneous tissue disorders) | 151/217 | 0/0 | 94/130 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Pain (Moderate) (Skin and subcutaneous tissue disorders) | 50/180 | 0/0 | 42/109 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Pain (Severe) (Skin and subcutaneous tissue disorders) | 5/166 | 0/0 | 6/90 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Redness (Any) (Skin and subcutaneous tissue disorders) | 30/137 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Redness (Mild) (Skin and subcutaneous tissue disorders) | 26/134 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 9/129 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Redness (Severe) (Skin and subcutaneous tissue disorders) | 2/127 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Swelling (Any) (Skin and subcutaneous tissue disorders) | 25/133 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 19/131 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 7/128 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Pain (Any) (Skin and subcutaneous tissue disorders) | 146/194 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Pain (Mild) (Skin and subcutaneous tissue disorders) | 129/184 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Pain (Moderate) (Skin and subcutaneous tissue disorders) | 49/148 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Pain (Severe) (Skin and subcutaneous tissue disorders) | 6/131 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Redness (Any) (Skin and subcutaneous tissue disorders) | 17/120 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Redness (Mild) (Skin and subcutaneous tissue disorders) | 13/118 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 6/117 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Redness (Severe) (Skin and subcutaneous tissue disorders) | 2/116 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Swelling (Any) (Skin and subcutaneous tissue disorders) | 18/121 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 15/120 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 5/117 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 1/115 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Pain (Any) (Skin and subcutaneous tissue disorders) | 127/175 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Pain (Mild) (Skin and subcutaneous tissue disorders) | 109/163 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Pain (Moderate) (Skin and subcutaneous tissue disorders) | 42/141 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Pain (Severe) (Skin and subcutaneous tissue disorders) | 5/117 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Fever >=38 degrees C (General disorders) | 13/169 | 0/0 | 17/96 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Fever >=38, <38.5 degrees C (General disorders) | 10/167 | 0/0 | 12/92 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Fever >=38.5, <39 degrees C (General disorders) | 2/165 | 0/0 | 5/90 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Fever >=39, =<40 degrees C (General disorders) | 3/167 | 0/0 | 2/87 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Fatigue (Any) (General disorders) | 119/204 | 0/0 | 86/128 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Fatigue (Mild) (General disorders) | 88/190 | 0/0 | 68/121 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Fatigue (Moderate) (General disorders) | 69/192 | 0/0 | 48/106 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Fatigue (Severe) (General disorders) | 20/173 | 0/0 | 12/93 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Headache (Any) (General disorders) | 84/189 | 0/0 | 53/114 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Headache (Mild) (General disorders) | 71/186 | 0/0 | 44/109 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Headache (Moderate) (General disorders) | 31/174 | 0/0 | 26/98 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Headache (Severe) (General disorders) | 4/167 | 0/0 | 6/90 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Vomiting (Any) (General disorders) | 36/173 | 0/0 | 5/89 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Vomiting (Mild) (General disorders) | 31/172 | 0/0 | 5/89 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Vomiting (Moderate) (General disorders) | 6/166 | 0/0 | 0/86 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Vomiting (Severe) (General disorders) | 2/165 | 0/0 | 0/86 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Diarrhea (Any) (General disorders) | 66/189 | 0/0 | 29/101 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Diarrhea (Mild) (General disorders) | 62/186 | 0/0 | 28/100 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Diarrhea (Moderate) (General disorders) | 14/171 | 0/0 | 3/87 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Diarrhea (Severe) (General disorders) | 5/168 | 0/0 | 1/87 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Muscle pain (Any) (General disorders) | 103/201 | 0/0 | 74/123 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Muscle pain (Mild) (General disorders) | 83/191 | 0/0 | 57/114 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Muscle pain (Moderate) (General disorders) | 46/183 | 0/0 | 31/99 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Muscle pain (Severe) (General disorders) | 9/168 | 0/0 | 7/91 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Joint pain (Any) (General disorders) | 48/181 | 0/0 | 31/99 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Joint pain (Mild) (General disorders) | 34/176 | 0/0 | 21/93 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Joint pain (Moderate) (General disorders) | 26/175 | 0/0 | 15/91 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Joint pain (Severe) (General disorders) | 5/167 | 0/0 | 4/90 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Fever >=38 degrees C (General disorders) | 13/131 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Fever >=38, <38.5 degrees C (General disorders) | 11/131 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Fever >=38.5, <39 degrees C (General disorders) | 3/126 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Fever >=39, =<40 degrees C (General disorders) | 3/126 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Fatigue (Any) (General disorders) | 98/171 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Fatigue (Mild) (General disorders) | 63/156 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Fatigue (Moderate) (General disorders) | 61/155 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Fatigue (Severe) (General disorders) | 13/131 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Headache (Any) (General disorders) | 53/152 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Headache (Mild) (General disorders) | 44/147 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Headache (Moderate) (General disorders) | 20/136 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Headache (Severe) (General disorders) | 2/128 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Vomiting (Any) (General disorders) | 20/135 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Vomiting (Mild) (General disorders) | 16/134 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Vomiting (Moderate) (General disorders) | 9/131 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Vomiting (Severe) (General disorders) | 1/126 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Diarrhea (Any) (General disorders) | 44/150 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Diarrhea (Mild) (General disorders) | 41/149 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Diarrhea (Moderate) (General disorders) | 13/134 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Diarrhea (Severe) (General disorders) | 2/127 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Muscle pain (Any) (General disorders) | 72/160 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Muscle pain (Mild) (General disorders) | 54/150 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Muscle pain (Moderate) (General disorders) | 40/143 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Muscle pain (Severe) (General disorders) | 8/131 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Joint pain (Any) (General disorders) | 37/147 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Joint pain (Mild) (General disorders) | 30/142 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Joint pain (Moderate) (General disorders) | 20/136 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Joint pain (Severe) (General disorders) | 3/129 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Fever >=38 degrees C (General disorders) | 8/120 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Fever >=38, <38.5 degrees C (General disorders) | 6/119 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Fever >=38.5, <39 degrees C (General disorders) | 4/117 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Fever >=39, =<40 degrees C (General disorders) | 2/116 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Fatigue (Any) (General disorders) | 77/157 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Fatigue (Mild) (Skin and subcutaneous tissue disorders) | 58/148 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Fatigue (Moderate) (General disorders) | 42/137 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Fatigue (Severe) (General disorders) | 8/120 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Headache (Any) (General disorders) | 53/142 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Headache (Mild) (General disorders) | 44/138 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Headache (Moderate) (General disorders) | 21/122 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Headache (Severe) (General disorders) | 4/119 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Vomiting (Any) (General disorders) | 13/120 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Vomiting (Mild) (General disorders) | 6/119 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Vomiting (Moderate) (General disorders) | 8/117 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Diarrhea (Any) (General disorders) | 30/130 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Diarrhea (Mild) (General disorders) | 26/128 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Diarrhea (Moderate) (General disorders) | 6/119 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Diarrhea (Severe) (General disorders) | 2/117 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Muscle pain (Any) (General disorders) | 61/152 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Muscle pain (Mild) (General disorders) | 47/142 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Muscle pain (Moderate) (General disorders) | 27/132 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Muscle pain (Severe) (General disorders) | 4/118 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Joint pain (Any) (General disorders) | 28/132 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Joint pain (Mild) (General disorders) | 23/128 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Joint pain (Moderate) (General disorders) | 13/122 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Joint pain (Severe) (General disorders) | 4/119 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 0/126 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Fever >40 degrees C (General disorders) | 0/165 | 0/0 | 0/86 | 0/0 | 0/0 — 13vPnC Dose 1 and Dose 4
Fever >40 degrees C (General disorders) | 0/126 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 2
Fever >40 degrees C (General disorders) | 0/115 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Vomiting (Severe) (General disorders) | 0/115 | 0/0 | 0/0 | 0/0 | 0/0 — 13vPnC Dose 3
Cholestasis (Hepatobiliary disorders) | 5 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.